CLINICAL TRIAL: NCT00518258
Title: Neuroimaging Studies of Depression in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Lee Blonder (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Lee Blonder, PI, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: R01-MH78228-2; R01MH078228 (NIH)
Record Dates: First submitted 2007-08-16; First posted 2007-08-20 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2013-04

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Magnetic Resonance Imaging (MRI); neuropsychological assessment
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patient Group
- 2: Control Group

SUMMARY:
The purpose of this study is to investigate similarities and differences in the neural pathways of depressed Parkinson's patients, non-depressed Parkinson's patients, and healthy controls using magnetic resonance imaging (MRI) of the brain and neuropsychological assessment.

DETAILED DESCRIPTION:
Depression is a common and potentially serious complication of Parkinson's disease (PD). Studies show that approximately 40 percent of PD patients are depressed. There is evidence that these patients have deficits in neuropsychological function relative to non-depressed PD patients. Despite the widespread toll on emotional health posed by PD, few studies have undertaken a comprehensive examination of the neural underpinnings of Parkinsonian depression. In this project, we will compare depressed versus non-depressed Parkinson patients to a sample of demographically-matched healthy controls using neuropsychological assessment and magnetic resonance imaging (MRI). To investigate possible effects of anti-Parkinsonian medication on mood, cognitive function, and neural response, PD patients will be tested both off and on Parkinsonian medications.

ELIGIBILITY:
Inclusion Criteria:

* right-handed
* willing/able to undergo magnetic resonance imaging (MRI)

Exclusion Criteria:

* history of neurological condition other than Parkinson's disease
* history of psychiatric condition other than depression
* history of substance abuse/dependence

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Neurology clinics, community sample
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2006-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee X. Blonder, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States